CLINICAL TRIAL: NCT05274061
Title: Couple's Retreats for PTSD: Healing the Impacts of Trauma in Texas Veteran Families
Brief Title: Couple's Retreats for Posttraumatic Stress Disorder
Acronym: PTSD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Nonrandomized, open-label study terminated at the end of the program's funding cycle.
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20210843H
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic stress disorder; Conjoint Therapy; Cognitive Behavioral Treatment; Intensive Treatments; Couples; Cognitive Behavioral Conjoint Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is an open-label, single group treatment study in which every couple will receive the intervention (AIM-CBCT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerated, Intensive, Multi-Couple Cognitive Behavioral Couples Therapy (AIM-CBCT for PTSD) (Experimental): This is a single-arm study in which each couple will receive AIM-CBCT. The intervention is described in the section below.
  Interventions: Behavioral: Accelerated, Intensive, Multi-Couple Cognitive Behavioral Couples Therapy

INTERVENTIONS:
Behavioral: Accelerated, Intensive, Multi-Couple Cognitive Behavioral Couples Therapy — AIM-CBCT consists of an accelerated, 2-day delivery of the first 7 sessions of CBCT for PTSD and is comprised of (a) psychoeducation about PTSD and relationship functioning; (b) instruction in conflict management skills; (c) instruction in effective communication skills with an emphasis on the identification and sharing of emotions to decrease emotional numbing and increase emotional intimacy; (d) discussion of the importance of approaching, rather than avoiding, difficult situations and identification of places, situations, people, and feelings that the couple has heretofore avoided as a result of PTSD; (e) instruction in identification of thoughts and related feelings that can maintain PTSD and relationship distress and strategies to increase cognitive flexibility, and (f) instruction in problem-solving skills to generate couple-level approach behaviors and guidance in how to select activities that double as opportunities to approach feared situations and engage in positive bonding.
  Other Names: AIM-CBCT for PTSD

SUMMARY:
Posttraumatic stress disorder (PTSD) increases the risk for conflict and dissatisfaction in romantic relationships. Accelerated, Intensive, Multi-Couples Cognitive Behavioral Conjoint Therapy (AIM-CBCT) is a behavioral treatment that targets reducing PTSD symptoms and improving relationship functioning. The treatment is delivered over two days using an intensive, outpatient group (between 2 to 6 couples) format. Previous research has found that AIM-CBCT for PTSD decrease PTSD symptoms and improves relationship functioning in military veterans and service members with combat-related PTSD. The present study examines whether these original findings can be replicated in a broader military/Veteran sample of up to 80 couples. The investigators predict that AIM-CBCT for PTSD will be associated with significant decreases in PTSD symptoms, depression, and anxiety in Veteran/military service members, significant decreases in mental health symptoms in their romantic partners, and an increase in couple's satisfaction for both the Veteran/service members and their partners.

Couples who agree to participate in the research study will be asked to participate in a 60-mintute pre-retreat meeting, the two-day retreat in which AIM-CBCT for PTSD will be delivered, and a 60-minute post-retreat check-in meeting. Additionally, each member of the couple will be asked to complete measures on their trauma history, mental health symptoms, and relationship functioning at baseline and at two and four weeks after the retreat.

DETAILED DESCRIPTION:
Numerous studies have documented an association between posttraumatic stress disorder (PTSD) symptoms and intimate relationship problems in Veterans and their partners, including relationship distress, physical and psychological aggression, and psychological distress in partners. Prior studies support the use of Cognitive-Behavioral Conjoint Therapy for PTSD (CBCT for PTSD) to treat PTSD and comorbid symptoms while simultaneously improving intimate relationship functioning. However, the standard outpatient format of CBCT for PTSD (i.e., fifteen 75-minute sessions over 15 weeks) presents challenges for many couples as well as for large-scale dissemination. To address these concerns, Dr. Steffany Fredman in collaboration with the STRONG STAR Consortium to Alleviate PTSD adapted CBCT for PTSD into an accelerated, intensive, multiple-couple format (AIM-CBCT for PTSD). The initial data of AIM-CBCT for PTSD tested in 24 couples was promising suggesting that this two-day retreat can reduce PTSD symptoms and improve mental health and relationship functioning in post-9/11 service members/veteran couples.

In September 2021, the South Texas Research Organizational Network Guiding Studies on Trauma and Resilience (STRONG STAR) initiated a clinical program which provides AIM-CBCT for PTSD to Texas Veteran couples impacted by PTSD symptoms. Within the clinical program, couples are asked to participate in an intake assessment to determine eligibility for treatment, a 60-minute pre-retreat meeting, a two-day retreat, a two-week post-retreat assessment, and a two-week post-retreat check-in. Couples who are eligible for the clinical program will be invited to participate in this replication study, which examines whether AIM-CBCT for PTSD is associated with reductions in PTSD and improvements in relationship functioning in a broader Veteran sample of up to 80 couples.

Research Questions and Hypotheses:

1. Will Accelerated, Intensive, Multi-Couple Cognitive Behavioral Couples Therapy delivered in a 2-day retreat (AIM-CBCT for PTSD) be associated with significant improvements in patient-rated PTSD symptom severity, as measured by the PTSD Checklist-DSM-5 (PCL-5), when assessed two-weeks and one month after treatment?

   Hypothesis 1: Participation in AIM-CBCT for PTSD will be associated with a significant reduction of self-reported PTSD symptoms on the Posttraumatic Checklist-DSM 5 (PCL-5) at the one-month follow-up assessment.
2. Will AIM-CBCT for PTSD be associated with significant improvements in secondary outcomes (e.g., patient self-reported comorbid symptom severity, relationship satisfaction) when assessed two-weeks and one month after treatment?

Hypothesis 2: Participation in AIM-CBCT for PTSD will be associated with a significant reduction of Veteran/Service members' self-reported mental health symptoms (Patient Health Questionnaire-9; General Anxiety Disorder-7) at the one-month follow-up assessment.

Hypothesis 3: Participation in AIM-CBCT for PTSD will be associated with a significant reduction of partners'' self-reported mental health symptoms (Patient Health Questionnaire-9; General Anxiety Disorder-7) at the one-month follow-up assessment.

Hypothesis 4: Participation in AIM-CBCT for PTSD will be associated with a significant increase in self-reported relationship satisfaction on the Couples Satisfaction Index-32) at the one-month follow-up assessment for both partners.

ELIGIBILITY:
Inclusion Criteria:

1. Cohabitating couples (ages 18 to 65 years old), who have been together for at least 4 months who reside in Texas.
2. At least one partner in the relationship is a Texas Veteran with significant PTSD symptoms as determined by the endorsement of at least one Criterion A event on the Life Event Checklist, the endorsement of at least one re-experiencing on the PCL-5 (i.e., a score of 2 or higher on Items 1, 2, 3, 4, or 5), the endorsement of at least one avoidance symptom on the PCL-5 (i.e., a score of 2 or higher on Items 6 or 7), and a total symptom score of 31 or higher on the PCL-5.
3. Both individuals must be willing to participate in the study.
4. Both individuals must be able to speak and read English.

Exclusion Criteria:

1. Couple is separated and/or is taking steps to dissolve their relationship (e.g., divorce).
2. Veteran or partner are currently participating in an evidence-based treatment for PTSD (Prolonged Exposure, Cognitive Processing Therapy, or Cognitive-Behavioral Conjoint Therapy for PTSD).
3. Veteran or partner exhibit current psychiatric symptoms warranting immediate intervention that is beyond the scope of the treatment provided in this study.
4. Veteran or partner exhibit evidence of a moderate or severe traumatic brain injury (as determined by the inability to comprehend the baseline screening questionnaires)
5. Veteran or partner report current suicidal ideation severe enough to warrant immediate attention (as determined by the Depressive Symptoms Index - Suicidality Subscale; DSI-SS)
6. Evidence or admission of severe intimate aggression as indicated by a "yes" endorsement to the one-question Screen for Conflict Question by Veteran or partner occurring within the past 6-months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist - DSM-5 (PCL-5) | Baseline, two-week post-retreat assessment, one-month post-retreat assessment
  Change in scale measurements by the PTSD CheckList-5. The PCL-5 is a 20-item, self-report measure of PTSD symptoms experienced in the past month. Each item is rated on a severity scale ranging from 0 (Not at all) to 4 (Extremely). The measure provides a total severity score that ranges from 0 to 80, with higher scores representing more PTSD symptoms.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline, two-week post-retreat assessment, one-month post-retreat assessment
  Change in scale measurements by the Patient Health Questionnaire-9. The PHQ-9 is 9-item, self-report screener for current depressive symptoms. Each item is rated on a frequency scale ranging from 0 (Not at all) to 3 (Nearly Every day). The measure provides a total severity score that ranges from 0 to 27, with higher scores representing more severe depressive symptoms.
General Anxiety Disorder - 7 (GAD-7) | Baseline, two-week post-retreat assessment, one-month post-retreat assessment
  Change in scale measurements by the Generalized Anxiety Disorder Screener: The GAD-7 is 7-item, self-report screener for current anxiety symptoms. Each item is rated on a frequency scale ranging from 0 (Not at all) to 3 (Nearly Every day). The measure provides a total severity score that ranges from 0 to 21, with higher scores representing more severe anxiety symptoms.
Couples Satisfaction Index-32 (CSI-32) | Baseline, two-week post-retreat assessment, one-month post-retreat assessment
  Change in scale measurements by the Couples' Satisfaction Index. The CSI-32 is 32-item, self-report measure of couple's satisfaction. Each item is rated on a 0 to 5 scale for a total score range of 0 to 161. Higher scores represent greater levels of relationship satisfaction with scores below 96 generally considered to reflect significant distress within the relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Alan L Peterson, PhD, Principal Investigator — UT Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fredman SJ, Le Y, Macdonald A, Monson CM, Rhoades GK, Dondanville KA, Blount TH, Hall-Clark BN, Fina BA, Mintz J, Litz BT, Young-McCaughan S, Jenkins AIC, Yarvis JS, Keane TM, Peterson AL; Consortium to Alleviate PTSD. A Closer Examination of Relational Outcomes from a Pilot Study of Abbreviated, Intensive, Multi-Couple Group Cognitive-Behavioral Conjoint Therapy for PTSD with Military Dyads. Fam Process. 2021 Sep;60(3):712-726. doi: 10.1111/famp.12654. Epub 2021 Apr 20. PMID 33876831
- [Background] Fredman SJ, Macdonald A, Monson CM, Dondanville KA, Blount TH, Hall-Clark BN, Fina BA, Mintz J, Litz BT, Young-McCaughan S, Hancock AK, Rhoades GK, Yarvis JS, Resick PA, Roache JD, Le Y, Wachen JS, Niles BL, McGeary CA, Keane TM, Peterson AL; Consortium to Alleviate PTSD. Intensive, Multi-Couple Group Therapy for PTSD: A Nonrandomized Pilot Study With Military and Veteran Dyads. Behav Ther. 2020 Sep;51(5):700-714. doi: 10.1016/j.beth.2019.10.003. Epub 2019 Nov 27. PMID 32800299
- [Background] Macdonald A, Fredman SJ, Taylor DJ, Pruiksma KE, Blount TH, Hall-Clark BN, Fina BA, Dondanville KA, Mintz J, Litz BT, Young-McCaughan S, Le Y, Jenkins AIC, Monson CM, Yarvis JS, Keane TM, Peterson AL; Consortium to Alleviate PTSD. Secondary individual outcomes following multicouple group therapy for posttraumatic stress disorder: An uncontrolled pilot study with military dyads. J Trauma Stress. 2022 Feb;35(1):321-329. doi: 10.1002/jts.22729. Epub 2021 Nov 20. PMID 34800060
- [Background] Monson CM, Taft CT, Fredman SJ. Military-related PTSD and intimate relationships: from description to theory-driven research and intervention development. Clin Psychol Rev. 2009 Dec;29(8):707-14. doi: 10.1016/j.cpr.2009.09.002. Epub 2009 Sep 10. PMID 19781836
- [Background] Monson CM, Fredman SJ. Cognitive-behavioral conjoint therapy for posttraumatic stress disorder: Harnessing the healing power of relationships. New York: Guilford. 2012
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841